CLINICAL TRIAL: NCT04153227
Title: Impact on Bone Health in Patients Undergoing Radical Cystectomy: Prevalence of Osteoporosis, Trabecular Bone Score (TBS) Assessment and Fracture Risk by FRAX in Male Patients After One Year of Radical Cystectomy
Brief Title: Osteoporosis, Trabecular Bone Score and Fracture Risk Assessment in Male Patients After Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Arturo Dominguez Garcia, Principal investigator, Parc Taulí Hospital Universitari
Other Study IDs: CEIm 2019/643
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Osteoporosis; Bladder Disease
Keywords: Osteoporosis; Trabecular bone score; FRAX; Radical cystectomy; Fracture risk; Metabolic acidosis; Vertebral fracture assessment; Bone mineral density; Urinary diversion
MeSH Terms: conditions — Osteoporosis; Urinary Bladder Diseases; Acidosis | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone mineral density (BMD) — Bone mineral density (BMD) is measured by Dual-energy X-ray absorptiometry (DXA). BMD provides a measure of bone mass.
Diagnostic Test: Trabecular bone score (TBS) — The Trabecular Bone Score (TBS) is a novel gray-level texture measurement that can be extracted from DXA images. TBS provides a measure of bone quality (bone microarchitecture).
Diagnostic Test: Fracture risk Assessment Tool (FRAX) — The Fracture risk Assessment Tool (FRAX) is a fracture risk calculator that estimates an individual's 10-year probability of incurring a hip or other major osteoporotic fracture.

SUMMARY:
Radical cystectomy (RC) with ileal urinary diversion (UD) is a standard treatment for muscle-invasive bladder cancer. However, emerging evidence indicates that this procedure may significantly impact bone health. Patients with UDs have a 21-48% higher risk of experiencing a fragility fracture compared to the general population. The underlying mechanisms are not entirely understood, but one prevailing hypothesis implicates substantial bone mineral density (BMD) loss due to the metabolic changes induced by UD, particularly driven by metabolic acidosis.

Dual-energy X-ray absorptiometry (DXA) remains the gold standard for measuring BMD and provides an indirect assessment of fracture risk. However, the trabecular bone score (TBS), a non-invasive imaging technique that evaluates bone microarchitecture, offers additional insights into bone quality that are independent of BMD and enhances the understanding of bone strength and fracture resistance. Furthermore, the use of tools such as the FRAX® (Fracture Risk Assessment Tool) helps in identifying patients at higher risk of osteoporotic fractures by estimating the 10-year probability of major fractures (MOF) (spine, forearm, hip, or shoulder) and hip fractures (HIP) based on various clinical risk factors. The predictive accuracy of FRAX® can be further refined by incorporating femoral neck BMD and adjusting for TBS.

Osteoporosis in men is a frequently underdiagnosed and undertreated condition. This underdiagnosis is also evident in patients with UDs. This study aims to evaluate the prevalence of bone alterations in men post-RC, employing both BMD and TBS measurements. Additionally, it seeks to identify key risk factors and critically assess the utility of FRAX® as a screening tool for pinpointing patients at elevated fracture risk.

To the best of the investigator's knowledge it will be the first study assessing the bone health after RC evaluating BMD, TBS and the fracture risk using the FRAX algorithm.

ELIGIBILITY:
Inclusion Criteria:

* All patients who understand, agree to participate and sign the informed consent.
* Males older than 50 years old.
* Patients undergoing radical cystectomy with ileal conduit or neobladder.
* Time over one year after radical cystectomy.

Exclusion Criteria:

* Female gender.
* Males below 50 years old.
* Radical cystectomy performed less than one year before.
* Radical cystectomy with cutaneous ureterostomy.
* Patients diagnosed with primary hyperparathyroidism.
* Patients receiving treatments that could influence bone metabolism, such as antiresorptive agents (including bisphosphonates or denosumab), chronic corticosteroids, androgen deprivation therapy for prostate cancer. Patients receiving treatment with Vitamin D were not excluded.
* Patients previously diagnosed with osteoporosis.
* Patients with a history of hemodialysis or renal transplantation.
* Patients receiving systemic cancer therapies for bladder tumor progression or other malignancies.
* Any patient who does not agree to participate or does not sign the informed consent

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males who underwent radical cystectomy with ileal urinary diversion (ileal conduit or neobladder).
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Bone mineral Density (BMD) | Baseline
  BMD values were categorized according to World Health Organization (WHO) criteria at any of the three measured sites: normal (T-score ≥ -1 SD), osteopenia (T-score between -1 and -2.5 SD), and osteoporosis (T-score ≤ -2.5 SD).

SECONDARY OUTCOMES:
Trabecular bone score (TBS) | Baseline
  Trabecular bone score (TBS) is a lumbar spine dual-energy absorptiometry texture index, which provides information on microarchitecture skeletal quality partially independent of BMD (TBS values >1.310 normal; TBS: 1.310-1.230 microarchitecture partially degraded; TBS <1.230 microarchitecture degraded).
Vertebral fractures | Baseline
  Presence of vertebral fractures evaluated by Vertebral Fracture Assessment (VFA)
Fracture Risk Assessment Tool (FRAX) | Baseline
  FRAX provides country-specific algorithms for estimating individualized 10-year probability of hip and major osteoporotic fracture (FRAX with and without BMD and FRAX with TBS). Criteria for starting antiresorptive treatment in Spain: Risk of major osteoporotic fracture at 10 years ≥7.5% (with BMD) or ≥10% (without BMD) or risk of hip fracture ≥3% (with or without BMD).

OTHER OUTCOMES:
Number of patients with metabolic acidosis. | Baseline
  Metabolic acidosis is considered if venous serum bicarbonate <22mmol/L
Number of patients with Secondary hyperparathyroidism. | Baseline
  Secondary hiperparathyroidism is considered if Serum parathyroid hormone (PTH) >65 pg/mL
Number of patients with Serum total 25(OH) vitamin D deficiency. | Baseline
  Serum total 25(OH) vitamine D deficiency is considered if <30 ng/mL
Number of patients with moderate-severe chronic kidney disease | Baseline
  Glomerular filtration rate (GFR) <60 mL/min

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Domínguez, MD, Principal Investigator — Hospital Universitari Parc Taulí
Locations (1):
- Hospital Universitari Parc Taulí, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: Undecided